CLINICAL TRIAL: NCT05678426
Title: TirolGESUND: General Exercise, Smoking Undone, and Nutrition Diet
Brief Title: TirolGESUND: Baseline-controlled Comparison of the Effects of Fasting Dietary Intervention or Smoking Cessation Combined With Exercise in Healthy Female Tyrolean Volunteers Aged 30-60 on Epigenetic and Multi-omic Biomarkers of Health, Ageing, and Disease
Acronym: TirolGESUND
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaet Innsbruck (Other)
Collaborators: Tirol Kiniken GmbH (Other)
Responsible Party: Principal Investigator, Martin Widschwendter, Study Coordinator/Co-Principal Investigator, Universitaet Innsbruck
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TirolGESUND; 20210420-2560 (Other: Studienregister des LKH - Universitätskliniken Innsbruck)
Record Dates: First submitted 2022-12-16; First posted 2023-01-10 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Healthy; Healthy Lifestyle; Smoking Cessation; Intermittent Fasting
Keywords: dna methylation; epigenetic age; intermittent fasting; smoking cessation; ketogenic supplement
MeSH Terms: conditions — Smoking Cessation; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoking cessation (Experimental): Smoking cessation encompasses three guided smoking cessation group therapy sessions (6-12 participants per session) followed by smoking cessation (occuring in the second session) for 6 months. Participants receive an optional exercise programme and motivational coaching over the duration of the study.
  Interventions: Behavioral: Smoking cessation
- Diet intervention (intermittent fasting) (Experimental): The dietary intervention encompasses induction (1 month) and maintenance (5 months) of a 16:8 intermittent fasting regime (time restricted eating to 8 h a day, fasting for remaining 16 h). During the introductory month, participants will only maintain a 14:10 intermittent fasting regime. Participants are randomized to receive a ketogenic supplement, medium-chain triglyceride fiber, to use daily. Participants receive an optional exercise programme and motivational coaching over the duration of the study.
  Interventions: Behavioral: Intermittent fasting; Behavioral: Intermittent fasting with ketogenic supplement

INTERVENTIONS:
Behavioral: Smoking cessation — Smoking cessation encompasses three guided smoking cessation group therapy sessions (6-12 participants per session) followed by smoking cessation (occuring in the second session) for 6 months. Participants receive an optional exercise programme and motivational coaching over the duration of the study.
  Arms: Smoking cessation
Behavioral: Intermittent fasting — The dietary intervention encompasses induction (1 month) and maintenance (5 months) of a 16:8 intermittent fasting regime (time restricted eating to 8 h a day, fasting for remaining 16 h). During the introductory month, participants will only maintain a 14:10 intermittent fasting regime. Participants receive an optional exercise programme and motivational coaching over the duration of the study.
  Arms: Diet intervention (intermittent fasting)
Behavioral: Intermittent fasting with ketogenic supplement — The dietary intervention encompasses induction (1 month) and maintenance (5 months) of a 16:8 intermittent fasting regime (time restricted eating to 8 h a day, fasting for remaining 16 h). During the introductory month, participants will only maintain a 14:10 intermittent fasting regime. Participants receive a ketogenic supplement, medium-chain triglyceride fiber, to use daily. Participants receive an optional exercise programme and motivational coaching over the duration of the study.
  Arms: Diet intervention (intermittent fasting)

SUMMARY:
The goal of this clinical study is to learn about disease-risk and age-associated changes in DNA methylation patterns associated with disease risk or age in healthy women aged 30-60 in response to health-promoting lifestyle intervention (intermittent fasting or smoking cessation). The main questions the study aims to answer are:

* Are the scores of DNA methylation in epigenetic signatures associated with age, women's cancer risk, or risk exposure reduced after 6 months of lifestyle intervention compared to baseline?
* What are the dynamics of DNA methylation changes during or following intervention, and do differences in changes between different sample types exist?
* Which other biomarkers of health and disease, including metabolic changes, microbiome, clinical, mental, or inflammatory parameters, are altered following intervention?

The investigators also aim to explore whether DNA methylation changes are associated with changes in other biomarkers mentioned above.

Participants will be allocated to intermittent fasting or smoking cessation based on inclusion criteria. Intermittent fasting encompasses a 16:8 intermittent fasting schedule. Food intake is limited to an 8 h window per day with fasting for the remaining 16 h. Within the intermittent fasting study, participants are randomised to receive a ketogenic supplement (medium-chain triglyceride fibre) or not. Participants in the smoking cessation study will be guided to stop smoking. All participants will receive 1:1 personal coaching throughout the study, and will be provided with an optional exercise programme. All participants will also receive nutritional advice from a professional dietician throughout the study. Participants are invited to donate samples every 2 months for 6 months.

Researchers will compare signatures at the start and after 6 months of intervention. Within the intermittent fasting group, researchers will compare effects in individuals that received the ketogenic supplement to those that did not.

DETAILED DESCRIPTION:
Background and study aims: A recent study reported that a majority of malignancies may be caused modifiable risk factors and could therefore be prevented. Smoking and diet are known risk factors for cancer but also other disorders such as cardiovascular or metabolic disorders and neurodegeneration, and may promote premature cellular ageing. The investigators and others have recently described epigenetic signatures for risk of being diagnosed, or developing future, women's cancers, as well as signatures reflecting cellular ageing and exposure to risk factors such as smoking. Utilization of DNA methylation biomarkers as surrogate endpoints indicative of current and/or future disease risk could improve future efforts in preventive medicine, both by providing information on disease risk and biofeedback. Few longitudinal studies have so far investigated the effects of lifestyle changes on DNA methylation and other biomarkers of health and disease.

TirolGESUND investigates the effect of two lifestyle interventions, smoking cessation or intermittent fasting (both with additional optional exercise), over 6 months for the promotion of health and reduction of disease risk, focusing on women's cancers.

Hypothesis: Intermittent fasting or smoking cessation for a duration of 6 months result in a modulation of scores of disease risk- and age-associated DNA methylation biomarker signatures in cervical samples, indicating a reduction of disease risk, exposure, or cellular ageing.

Study design: TirolGESUND is a baseline-controlled intervention study with two parallel arms, smoking cessation and intermittent fasting. Participants are allocated to the study arm based on eligibility criteria. Within the intermittent fasting arm, participants are randomised to receive a ketogenic supplement or not. Ketosis has been suggested to elicit beneficial metabolic alterations and could therefore further enhance beneficial effects in the dietary intervention.

Endpoints: The primary endpoint are score changes in epigenetic biomarkers of cellular ageing and disease risk, primarily recently published Women's cancer risk identification (WID) indices.

In secondary and subsidiary outcomes, the study will explore temporal and spatial dynamics of DNA methylation alterations in response to lifestyle interventions, comparing different surrogate samples (blood, buccal, cervical).

The study also investigates the impact of lifestyle intervention on other biomarkers of health and disease as a pilot study for future behavioural studies in the space of disease prevention and ageing research.

Intervention: Participants will be allocated to intermittent fasting or smoking cessation based on inclusion criteria. Intermittent fasting encompasses a 16:8 intermittent fasting schedule. Food intake is limited to an 8 h window per day with fasting for the remaining 16 h. Within the intermittent fasting study, participants are randomised to receive a ketogenic supplement (medium-chain triglyceride fibre) or not. Participants in the smoking cessation study will be guided to stop smoking. All participants will receive 1:1 personal coaching throughout the study, and will be provided with an optional exercise programme. All participants will also receive nutritional advice from a professional dietician throughout the study.

The duration of the study including intervention is 6 months for each participant. Participants are invited to return for optional sample collection visits at 12 and 18 months.

Visits and examinations: The following samples will be collected at baseline and subsequently every two months for 6 months: cervical, buccal, blood, fecal, urine and saliva samples. At the beginning and end of the study, participants will additionally receive sports medicine examinations (spirometry, ergometry/sports medicine exam) and an examination of vascular health. Participants are asked to complete an epidemiological questionnaire at the beginning of the study and receive additional questionnaires throughout the study to monitor food intake (prior to every visit), physical activity (once a month), or quality of life (baseline, 6 months). Participants may optionally donate skin biopsies at baseline and after 6 months.

Participants receive a fitness tracker to monitor physical activity and exercise in an objective manner. Some participants in the intermittent fasting group are receiving a capillary blood monitor to evaluate ketosis levels at the end of the fasting period three times a week.

Randomization in the intermittent fasting study arm: Participants are randomised to receive or to not receive ketogenic supplement 1:1 using menopause- and BMI-stratified block randomization.

Participant risks and benefits: Participants will receive support in implementing (putative) health-promoting interventions, including giving up smoking and intermittent fasting over 6 months, and are hence expected to personally benefit from participation. Risks are expected to be minimal as the study involves only a behavioural/lifestyle change, but can include e.g. development of haematoma after blood sampling, mood swings due to smoking cessation, or hunger at the initiation of intermittent fasting.

Sample size: Dynamics of DNA methylation changes are unknown at the start of the study, rendering sample size estimation challenging. For each study arm (intermittent fasting, intermittent fasting plus ketogenic supplement, smoking cessation) n=60 participants are recruited based on prior information of standard deviation in DNA methylation indices.

Expected Drop-Out levels: Based on prior literature in lifestyle or dietary interventions, drop-out rates of 15-20% are expected.

Data management and protection: Clinical data is recorded using an electronic case report form with validity checks. Laboratory data is analysed in a coded manner. Data protection follows the principles of the European General Data Protection Regulation (GDPR).

Quality control: Standard operating procedures for sample collection and clinical procedures have been designed and implemented.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 30 to 60
2. Motivated to change their lifestyle

Smoking cessation intervention:

3a. Smoking cessation: ≥10 cigarettes per day for at least the last five years

Dietary intervention:

3b Dietary intervention: BMI between 25 and 35

NB [Nota Bene], should 3a and 3b apply, participant will be allocated to the smoking cessation intervention.

Exclusion Criteria:

1. Relevant underlying conditions:

   1. Current or previous malignant tumour or cancer
   2. Current or previous significant cardiovascular disorder [participants with elevated blood pressure are allowed to participate as long as it is well controlled under their current medication]
   3. Current or previous metabolic disorder (e.g., diabetes type I or II) [in the dietary intervention arm, participants with current hypothyroidism/Morbus Hashimoto will be excluded as the switch to intermittent fasting may require a adjustment of their medication]
   4. Current or previous psychiatric disorder (e.g., eating disorder, depression)
2. Current pregnancy or lactation period
3. Total hysterectomy
4. Known current or previous premalignant lesion of the cervix uteri (CIN2/3)
5. Concurrent participation in another interventional trial

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline scores of DNA methylation biomarkers of age, disease risk, and exposure | Baseline, Month 6 (per participant)
  Examination of change in epigenetic age, disease risk, and exposure signature scores compared to baseline (before and after intervention, i.e. baseline-controlled) in cervical samples. DNA methylation levels will be measured using the Illumina MethylationEPIC array and computed using previously described methylation indices, including:
  * WID-BC (Women's risk identification - Breast cancer)
  * WID-OC (ovarian cancer)
  * WID-EC (endometrial cancer)
  * WID-CIN (cervical intraepithelial neoplasia)
  * WID-REA (relative epithelial age)
  * WID-RIA (relative immune age)
  * pcgtAge (mitotic clock)
  * WID-SOLA[ge] (systemic organ life age)
  * WID-SMK (smoking)

SECONDARY OUTCOMES:
Description of study characteristics: registration rate in percent (%) | Baseline
  Final registration rate of participants initially interested, i.e. those who signed up for information webinars, in percent (%)
Description of study characteristics: drop-out rate in percent (%) | Month 6 (Primary end point of study)
  Number of included participants who dropped out over the course of the study, in percent (%)
Description of study characteristics: compliance rate in percent (%) | Month 6 (Primary end point of study)
  Description of compliance rate (i.e. days compliant with the intervention over the duration of the study), in percent (%)
Change in DNA methylation scores from baseline in cervical samples at month 2, month 4, and month 6 | Samples collected at baseline, month 2, month 4, and month 6
  Examination of change in epigenetic age, disease risk, and exposure signature scores compared to baseline (before and after intervention, i.e. baseline-controlled) in cervical samples collected at baseline and again at month 2, 4, and 6, using t Tests and/or linear mixed-effects models where appropriate. DNA methylation levels will be measured using the Illumina MethylationEPIC array and computed using previously described methylation indices, including:
  * WID-BC
  * WID-OC
  * WID-EC
  * WID-CIN
  * WID-REA (relative epithelial age)
  * WID-RIA (relative immune age)
  * pcgtAge (mitotic clock)
  * WID-SOLA[ge]
  * WID-SMK
  The change in scores will also be compared to changes in the same scores in buccal and blood samples (outcomes 6 and 7) to evaluate temporal and spatial DNA methylation dynamics in response to lifestyle intervention.
Change in DNA methylation scores from baseline in buccal samples at month 2, month 4, and month 6 | Samples collected at baseline, month 2, month 4, and month 6
  Examination of change in epigenetic age, disease risk, and exposure signature scores compared to baseline (before and after intervention, i.e. baseline-controlled) in buccal samples collected at baseline and again at month 2, 4, and 6, using t Tests and/or linear mixed-effects models where appropriate. DNA methylation levels will be measured using the Illumina MethylationEPIC array and computed using previously described methylation indices, including:
  * WID-BC
  * WID-OC
  * WID-EC
  * WID-CIN
  * WID-REA (relative epithelial age)
  * WID-RIA (relative immune age)
  * pcgtAge (mitotic clock)
  * WID-SOLA[ge]
  * WID-SMK
  The change in scores will also be compared to changes in the same scores in cervical and blood samples (outcomes 5 and 7) to evaluate temporal and spatial DNA methylation dynamics in response to lifestyle intervention.
Change in DNA methylation scores from baseline in blood samples at month 2, month 4, and month 6 | Samples collected at baseline, month 2, month 4, and month 6
  Examination of change in epigenetic age, disease risk, and exposure signature scores compared to baseline (before and after intervention, i.e. baseline-controlled) in blood samples collected at baseline and again at month 2, 4, and 6, using t Tests and/or linear mixed-effects models where appropriate. DNA methylation levels will be measured using the Illumina MethylationEPIC array and computed using previously described methylation indices, including:
  * WID-BC
  * WID-OC
  * WID-EC
  * WID-CIN
  * WID-REA (relative epithelial age)
  * WID-RIA (relative immune age)
  * pcgtAge (mitotic clock)
  * WID-SOLA[ge]
  * WID-SMK
  The change in scores will also be compared to changes in the same scores in cervical and buccal samples (outcomes 5 and 6) to evaluate temporal and spatial DNA methylation dynamics in response to lifestyle intervention.
Change in beneficial and harmful microbial species compared to baseline, in percent (%) | Samples collected at baseline and month 6, optional month 2 and month 4
  Quantification of selected beneficial and harmful bacteria based on previous literature, in fecal and saliva samples, and computation of change from baseline.
  If big differences are found, temporal dynamics of changes will be examined in samples collected at month 2 and month 4.
Change in microbial diversity score compared to baseline, in percent (%) | Samples collected at baseline and month 6, optional month 2 and month 4
  Quantification of microbial diversity using entropy scores at baseline and month 6. If big differences are found, temporal dynamics of changes will be examined in samples collected at month 2 and month 4.
Change of immune and inflammatory cell populations in peripheral blood | Samples collected at baseline and month 6, optional month 2 and month 4
  Immune/inflammatory cell heterogeneity will be investigated in samples from peripheral blood using flow cytometry using well-established cellular markers. Cell population changes from baseline will be reported. If big differences are found, temporal dynamics of changes will be examined in samples collected at month 2 and month 4. Pending the outcome of this investigation, targeted investigation of associated plasma circulating markers may be conducted.
Change in body mass index from baseline | Baseline and month 6.
  Changes in BMI from baseline (diet arm of the study).
  Changes in BMI from baseline (diet arm of the study).
Change in body composition as quantified by bioelectric impedance analysis from baseline | Baseline and month 6.
  Change in body composition (% muscle, fat, water, abdominal fat composition) composition from baseline as quantified by bioelectric impedance analysis (diet arm of the study).
Change in smoking status from baseline | Baseline and month 6.
  Changes in smoking status (smoking cessation arm of the study), defined as: smoking - yes/no.
Change in vascular health from baseline: pulse-wave velocity | Baseline and month 6.
  Change in measured pulse wave velocity (m/s) as recorded using the vicorder.
Change in vascular health from baseline: intima-media thickness | Baseline and month 6.
  Change in measured vascular intima-media thickness as measured using ultrasound.
Change in vascular health from baseline: intima-media thickness | Baseline and month 6.
  Change in measured vascular plaque score as measured using ultrasound.
Change in physical activity from baseline | Baseline and month 6
  Change in physical activity from baseline, as quantified using the international physical activity questionnaire (IPAQ)
Change in physical activity from baseline: fitness tracker data | Baseline and month 6
  Change in physical activity from baseline as quantified using fitness tracker data (resting heart rate month 0 to resting heart rate month 6)
Change in physical activity from baseline: VO2max | Baseline and month 6
  Change in physical activity from baseline as quantified via sports examination (VO2max)
Change in pulmonary health from baseline | Baseline and month 6
  Pulmonary health markers, e.g. FEV1 (Forced expiratory volume), at baseline and at 6 months using spirometry
Change in health-related quality of life from baseline | Baseline and month 6
  Change in health-related quality of life (EuroQoL, i.e. EQ-5D-5L, https://euroqol.org/eq-5d-instruments/eq-5d-5l-about/) at baseline and at 6 months

OTHER OUTCOMES:
Exploratory investigation of metabolic profile via NMR over course of intervention for hypothesis generation | Urine and saliva samples collected at baseline, month 2, month 4, and month 6
  The investigators will examine metabolome profiles in urine and saliva samples using untargeted nuclear magnetic resonance (NMR) for hypothesis generation of future intervention trials.
Change of plasma inflammatory markers compared to baseline. | Samples collected at baseline and month 6, optional month 2 and month 4
  Pending the outcome of this investigation, targeted investigation of associated plasma circulating markers may be conducted. Appropriate inflammatory markers will be investigated using a sufficiently sensitive method, such as high sensitivity ELISA or luminex bead arrays.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Widschwendter, MD, Principal Investigator — Universitaet Innsbruck
Locations (1):
- European Translational Oncology Prevention and Screening Institute, Hall in Tirol, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study, in particular epigenetic, metabolomic, and microbial will be stored in a publicly available but access-controlled repository (EGA-European Genome Phenome Archive, https://ega-archive.org/, or similar), due to the sensitive nature of epigenetic data. All data will only be shared in a coded (pseudonymised) or completely anonymised format. Prior to use, any potential collaborators must sign a data access agreement and comply with the terms of data sharing.
  Some datasets (summary characteristics, or completely anonymised results) may additionally be published as a supplement to the results publications.
Supporting Information: SAP, CSR, Analytic Code
Time Frame: Data will be deposited when summary data are published.
Access Criteria: Data will be restricted for non-commercial research in the space of healthy ageing research. Sharing is restricted to certain geographical areas that have high GDPR standards.

REFERENCES:
- [Background] GBD 2019 Cancer Risk Factors Collaborators. The global burden of cancer attributable to risk factors, 2010-19: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2022 Aug 20;400(10352):563-591. doi: 10.1016/S0140-6736(22)01438-6. PMID 35988567
- [Background] Jacob L, Freyn M, Kalder M, Dinas K, Kostev K. Impact of tobacco smoking on the risk of developing 25 different cancers in the UK: a retrospective study of 422,010 patients followed for up to 30 years. Oncotarget. 2018 Apr 3;9(25):17420-17429. doi: 10.18632/oncotarget.24724. eCollection 2018 Apr 3. PMID 29707117
- [Background] Key TJ, Allen NE, Spencer EA, Travis RC. The effect of diet on risk of cancer. Lancet. 2002 Sep 14;360(9336):861-8. doi: 10.1016/S0140-6736(02)09958-0. PMID 12243933
- [Background] Steck SE, Murphy EA. Dietary patterns and cancer risk. Nat Rev Cancer. 2020 Feb;20(2):125-138. doi: 10.1038/s41568-019-0227-4. Epub 2019 Dec 17. PMID 31848467
- [Background] Barrett JE, Herzog C, Jones A, Leavy OC, Evans I, Knapp S, Reisel D, Nazarenko T, Kim YN, Franchi D, Ryan A, Franks J, Bjorge L, Zikan M, Cibula D, Harbeck N, Colombo N, Dudbridge F, Jones L, Sundstrom K, Dillner J, Radestad AF, Gemzell-Danielsson K, Pashayan N, Widschwendter M. The WID-BC-index identifies women with primary poor prognostic breast cancer based on DNA methylation in cervical samples. Nat Commun. 2022 Feb 1;13(1):449. doi: 10.1038/s41467-021-27918-w. PMID 35105882
- [Background] Barrett JE, Sundstrom K, Jones A, Evans I, Wang J, Herzog C, Dillner J, Widschwendter M. The WID-CIN test identifies women with, and at risk of, cervical intraepithelial neoplasia grade 3 and invasive cervical cancer. Genome Med. 2022 Oct 19;14(1):116. doi: 10.1186/s13073-022-01116-9. PMID 36258199
- [Background] Barrett JE, Jones A, Evans I, Reisel D, Herzog C, Chindera K, Kristiansen M, Leavy OC, Manchanda R, Bjorge L, Zikan M, Cibula D, Widschwendter M. The DNA methylome of cervical cells can predict the presence of ovarian cancer. Nat Commun. 2022 Feb 1;13(1):448. doi: 10.1038/s41467-021-26615-y. PMID 35105887
- [Background] Barrett JE, Herzog C, Kim YN, Bartlett TE, Jones A, Evans I, Cibula D, Zikan M, Bjorge L, Harbeck N, Colombo N, Howell SJ, Radestad AF, Gemzell-Danielsson K, Widschwendter M. Susceptibility to hormone-mediated cancer is reflected by different tick rates of the epithelial and general epigenetic clock. Genome Biol. 2022 Feb 22;23(1):52. doi: 10.1186/s13059-022-02603-3. PMID 35189945